CLINICAL TRIAL: NCT07350798
Title: Applicability of Robotic Devices, Virtual and Augmented Reality in the Rehabilitation of People With Stroke During Treadmill Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Head of Department, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IG/1357-0/2025
Record Dates: First submitted 2025-12-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: stroke; robotic; virtual reality; augmented reality; rehabilitation; treadmill training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TT (Experimental): Receiving high intensity treadmill training
  Interventions: Other: Treadmill Training
- R-TT (Experimental): Receiving high intensity treadmill training with ReStore robotic device.
  Interventions: Other: Robot Assisted Treadmill Training
- VR&AR-TT (Experimental): Receiving treadmill training with C-Mill, a special treadmill that provides virtual and augmented reality.
  Interventions: Other: Treadmill Training with Virtual and Augmented Reality
- C-TT (Experimental): Receiving treadmill training with the combination of the ReStore and C-Mill system.
  Interventions: Other: Combined Treadmill Training

INTERVENTIONS:
Other: Treadmill Training — The TT group performs high-intensity treadmill training on a conventional treadmill. 5 times/week for 3 weeks, 30 minutes each.
  Arms: TT
Other: Robot Assisted Treadmill Training — The TT group performs high-intensity treadmill training on a conventional treadmill. Before the training begins, the ReStore Soft exoskeleton, which is a special gait assist device, is fitted. The device uses motion sensors to process the movements of the lower limb on the healthy side and uses a motor attached to the waist to map them using bowden cables while walking on the affected paretic side in real time. During therapy, the amount of assistance provided by the exoskeleton can be continuously adjusted to the patient's needs from an external controller, so that therapy can be performed in a specialized manner for the individual. 5 times/week for 3 weeks, 30 minutes each.
  Arms: R-TT
Other: Treadmill Training with Virtual and Augmented Reality — The VR&AR-TT group performs treadmill training on a special treadmill, the C-Mill VR+ device, for which the virtual and augmented reality movement programs are provided by the CueFors 2.5 software, which is the original control software for the C-Mill. The C-Mill VR+ system is a 3 m long and 1 m wide treadmill with a force platform underneath. A 65" fixed-position monitor in front of the treadmill provides the virtual reality environment, and a projector placed next to the treadmill allows various tasks to be projected onto the treadmill belt, providing immediate real-time feedback to the patient and therapist via the force platform. 5 times/week for 3 weeks, 30 minutes each.
  Arms: VR&AR-TT
Other: Combined Treadmill Training — Patients in the C-TT group use the ReStore Soft exoskeleton and the C-Mill VR+ system together. 5 times/week for 3 weeks, 30 minutes each.
  Arms: C-TT

SUMMARY:
* Objective assessment of clinical symptoms, mobility and quality of life changes resulting from stroke and determination of changes resulting from therapies.
* Assessment of the rehabilitation effectiveness of traditional treadmill training.
* Assessment of the rehabilitation effectiveness of gait training performed on a treadmill with a robot-assisted soft-exoskeleton.
* Assessment of the rehabilitation effectiveness of treadmill training supplemented with virtual and augmented reality.
* Determination of the joint application possibilities of robot-assisted and virtual and augmented reality treadmill training in order to further increase the effectiveness.
* Comparison of the effectiveness of different treadmill trainings.
* Mapping of changes in gait patterns due to therapies using 3D motion analysis.
* Mapping of changes in postural stability due to therapies using posturography.

ELIGIBILITY:
Inclusion Criteria:

* has had a first ischemic stroke diagnosed by a neurologist based on CT or MRI;
* neurological examination shows mobility and postural limitations;
* mRS score of 2 or higher;

Exclusion Criteria:

* multiple strokes in the medical history;
* systolic blood pressure less than 120 or greater than 160 mmHg;
* orthostatic hypotension;
* carotid artery stenosis;
* severe heart disease;
* hemophilia;
* traumatic brain injury;
* seizure disorder; untreated diabetes;
* abnormal electroencephalography;
* Mini Mental Test score < 22;
* abnormal blood panel;
* use of sedatives; irregular medication;
* severe aphasia (Western Aphasia Battery ≤ 25);
* severe vision or hearing impairment;
* severe sensory dysfunction;
* severe orthopedic problem;
* other neurological condition affecting motor function;
* alcoholism;
* drug use;
* smoking after stroke diagnosis;
* inability to walk at least 100 m with or without assistive devices in 6 minutes;
* BBS score ≤ 32;
* BI score ≤ 70;
* inability to understand verbal instructions or signals on a television screen;
* current participation in an individual or group exercise program outside of standard physiotherapy;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 3 weeks
  The modified Rankin Scale (mRS) indicates the degree of independence in daily activities and the severity of disability. The method for assessing mRs is a guided interview. . The scoring is divided as follows: 0-No symptoms; 1-No significant disability. Able to carry out activities of daily living despite some symptoms; 2-Mild disability. Able to look after himself without assistance but not able to carry out all previous activities; 3-Moderate disability. Needs some assistance with activities of daily living but can walk without assistance; 4-Moderately severe disability. Unassisted, unable to meet his/her own physical needs, unable to walk without assistance; 5-Severe disability. Bedridden, incontinent, requires constant nursing care; 6-Dead

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) | 3 weeks
  The SF-36 (36-Item Short Form Health Survey) is a widely used, patient-reported questionnaire that assesses health-related quality of life across 8 domains: physical functioning, bodily pain, role limitations (physical & emotional), vitality, social functioning, mental health, and general health perceptions. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table.The scores from those questions that address each specific area of functional health status are then averaged together, for a final score within each of the 8 dimensions measured. (eg pain, physical functioning etc.)
Stroke Impact Scale-16 (SIS-16) | 3 weeks
  The Stroke Impact Scale-16 (SIS-16) consists of 16 items from the 4 physical domains (strength, hand function, mobility, and ADL/IADL). Scoring involves rating 16 physical function items on a 1-to-5 Likert scale (1=could not do at all, 5=not difficult at all), with higher scores indicating better function.
Berg Balance Scale (BBS) | 3 weeks
  The Berg Balance Scale (BBS) was used to measure static and dynamic balance. The BBS can objectively measure the subject's ability to balance safely during a series of pre-determined tasks. It is a 14-item task, with each item scored on a five-point scale from 0 to 4, where 0 indicates the lowest level of function and 4 the highest. The maximum score is 56, indicating perfect functional balance. A score below 45 indicates an increased risk of falling, and, the lower the score, the higher the risk of falling.
Tinetti test | 3 weeks
  The Tinetti test is a common clinical tool for assessing mobility, balance (static and dynamic) and gait in the elderly, especially for assessing fall risk. Scoring: 0, 1, 2 points for each subscale. Total score 28. A score below 25 points significantly increases the likelihood of falling
6 minute walking test (6MWT) | 3 weeks
  To measure endurance, we used a 6-minute walk test (6mWT). During the test, the subject walks back and forth along a pre-designated flat and straight 50 m long trail. The walk starts when the timer is started at the tester's command; the pace of the walk is set by the subject, with no interference from the tester. If the subject needs to stop for a rest during the walk, the timing is not stopped. The subject will continue walking for 6 min and will stop only at the direction of the examiner after the 6 min have elapsed. The result is the distance covered in 6 min, expressed in meters. If the subject is required to stop and sit down within the 6 min, the test result is the distance covered. The greater the distance traveled, the better the endurance required.
10 meter walking test | 3 weeks
  A 10-meter walk test (10mWT) was used to measure walking speed. To perform the test, a 10 m long flat, level area was designated. The 10 m section was marked at 0, 2, 8 and 10 m with thick adhesive tape. The subject started walking at the 0 m mark on the instructions of the examiner. As soon as he reached the 2 m mark, the examiner started the timer and stopped it the moment he reached the 8 m mark, thus testing his walking speed over a 6 m stretch. The speed is given by the distance (6 m) divided by the time measured (in seconds to two decimal places) in m/s
Posturographic examination | 3 weeks
  During the postural examination, the presence and extent of postural instability were monitored using a posturograph (ProKin 252N, TecnoBody, Dalmine, Italy). During the test, the subjects were asked to stand on the test apparatus for 20 s in 4 different in-creasingly difficult postures: 1-wide stance-eye open (WEO); 2-wide stance-eye closed (WEC); 3-narrow stance-eye open (NEO); 4-narrow stance-eye closed (NEC). During the test, the subjects stood barefoot on the test apparatus and were not exposed to any external stimuli during the test. The results are provided by the 3-dimensional path of the body's center of pressure (COP-Sway). The smaller the COP-Sway , the lower the postural instability.
3D gait analysis - Spatiotemporal parameters | 3 weeks
  For 3D gait analysis we use the MVN Awinda motion capture system developed by Xsens (Movella, El Segundo, Califonia, US) and the MVN Analyze (version 2025.0.1.) motion analysis software. The MVN Awinda motion capture system consists of a total of 17 inertial measurement units (IMUs), which include accelerometers, gyroscopes, and magnetometers. The sensors are placed at different predefined anatomical points on the body.
  The 3D gait analysis includes multiple distinct gait parameters, each representing an independent outcome with its own unit of measure. These parameters are not aggregated into a single composite score, but are analyzed and reported separately as standard spatiotemporal gait outcomes.
  Spatiotemporal parameters: Gait speed (m/s); Number of steps (count); Cadence (steps/min).
3D gait analysis - Spatial parameters | 3 weeks
  For 3D gait analysis we use the MVN Awinda motion capture system developed by Xsens (Movella, El Segundo, Califonia, US) and the MVN Analyze (version 2025.0.1.) motion analysis software. The MVN Awinda motion capture system consists of a total of 17 inertial measurement units (IMUs), which include accelerometers, gyroscopes, and magnetometers. The sensors are placed at different predefined anatomical points on the body.
  The 3D gait analysis includes multiple distinct gait parameters, each representing an independent outcome with its own unit of measure. These parameters are not aggregated into a single composite score, but are analyzed and reported separately as standard spatiotemporal gait outcomes. Spatial parameters: Step length - Left (cm); Step length - Right (cm); Step length difference (cm); Step width - Left (cm); Step width - Right (cm); Step width difference (cm).
10. 3D gait analysis - Temporal parameters | 3 weeks
  For 3D gait analysis we use the MVN Awinda motion capture system developed by Xsens (Movella, El Segundo, Califonia, US) and the MVN Analyze (version 2025.0.1.) motion analysis software. The MVN Awinda motion capture system consists of a total of 17 inertial measurement units (IMUs), which include accelerometers, gyroscopes, and magnetometers. The sensors are placed at different predefined anatomical points on the body. The 3D gait analysis includes multiple distinct gait parameters, each representing an independent outcome with its own unit of measure. These parameters are not aggregated into a single composite score, but are analyzed and reported separately as standard spatiotemporal gait outcomes. Temporal parameters (percentage of gait cycle): Total gait cycle - Left (%); Total gait cycle - Right (%); Swing phase - Left (%); Swing phase - Right (%); Stance phase - Left (%); Stance phase - Right (%); Double support phase - Left (%); Double support phase - Right (%).

CONTACTS AND LOCATIONS:
Overall Officials: József Dr. habil. Tollár, Principal Investigator — Somogy County Kaposi Mór Teaching Hospital
Locations (1):
- Somogy County Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No